CLINICAL TRIAL: NCT03754465
Title: A Phase 2 Clinical Study to Evaluate the Efficacy and Safety of ALLO-ASC-SHEET in Subjects with Diabetic Foot Ulcers
Brief Title: Clinical Study of ALLO-ASC-SHEET in Subjects with Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLO-ASC-SHEET-102
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALLO-ASC-DFU (Experimental): Experimental: ALLO-ASC-DFU Hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-DFU
- Hydrogel SHEET(Vehicle control) (Placebo Comparator): Placebo Comparator: Vehicle Control Hydrogel sheet without allogenic adipose-derived mesenchymal stem cells
  Interventions: Procedure: Hydrogel SHEET(Vehicle control)

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU Sheet to diabetic foot ulcer
  Other Names: Hydrogel sheet containing Allogenic Mesenchymal Stem Cells
  Arms: ALLO-ASC-DFU
Procedure: Hydrogel SHEET(Vehicle control) — Application of Hydrogel SHEET to diabetic foot ulcer
  Other Names: Hydrogel sheet without Allogenic Mesenchymal Stem Cells
  Arms: Hydrogel SHEET(Vehicle control)

SUMMARY:
This is a phase 2 double-blind clinical study to evaluate the efficacy and Safety of ALLO-ASC-SHEET in subjects with Diabetic Foot Ulcers, compared to placebo therapy.

DETAILED DESCRIPTION:
1. Active Group: ALLO-ASC-SHEET
2. Control Group: Hydrogel SHEET (vehicle control)
3. Study Type: Interventional
4. Study Design: Randomized, Comparator-controlled, Double-blind, multi-center study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 18 and 80 years of age.
2. Diagnosed with Type I or Type II diabetics and has diabetic foot ulcers for longer than 4 weeks at the screening visit.
3. Foot ulcer located in the instep, border or sole of the foot, with ulcer size between 1 cm2 and 15 cm2.
4. Ulcer graded I by Wagner grade, and extended to skin, subcutaneous tissue, but without exposure of muscle, tendon, bone or joint capsule.
5. Ulcer is free of necrotic debris, exhibits no signs of clinical infection.
6. Ulcer area blood circulation meets one of the following criteria

   * A. Blood vessels around the ulcer detected by Doppler Test
   * B. range of Ankle Brachial Index(ABI) was > 0.7 to < 1.3
   * C. Transcutaneous oxygen pressure, (TcPO2) > 30 mmHg.
7. Is able to give written informed consent prior to study start and to comply with the study requirements.

Exclusion Criteria:

1. Ulcer is of non-diabetic pathophysiology.
2. The ulcer has increased or decreased in size by ≥ 30% during the week after the Screening Visit.
3. Is Human Immunodeficiency Virus (HIV) positive?
4. Have severe hepatic deficiencies.
5. Have a glycated hemoglobin A1c (HbA1c) level of > 10%.
6. Have allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue.
7. Require intravenous (IV) antibiotics to treat the target wound infection.
8. Have severe renal failure including subject on renal dialysis.
9. Pregnant or breast-feeding.
10. Is unwilling to use an "effective" method of contraception during the study.
11. Have evidence of current infection including pus drainage from the wound site.
12. Have a clinically relevant history of alcohol or drugs abuse.
13. Have postprandial blood sugar > 350 mg/dl.
14. Is not able to understand the objective of this study or to comply with the study requirements.
15. Is considered by the investigator to have a significant disease which might have impacted the study.
16. Is considered not suitable for the study by investigator.
17. Have a history of malignancy within the last five years (except basal cell carcinoam in situ).
18. Is currently or were enrolled in another clinical study within 60 days of screening.
19. Have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days.
20. Is receiving oral or parenteral corticosteroids, immunosuppressive, or cytotoxic agents with unstable dose prior to 4 weeks from screening.
21. Cannot maintain off-loading process
22. Panel reactive antibody (PRA) levels ≥ 20%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Proportions of subjects who achieved complete wound closure | During 12 weeks
  Proportions of subjects who achieved complete wound closure

SECONDARY OUTCOMES:
Time to initial complete wound closure between the two groups | During 12 weeks
  Time to initial complete wound closure between the two groups
Changes in wound size compared to baseline between the two groups | During 12 weeks
  Wound size is measured by using eKare 3D Wound Measurement system(Mobile Devices)
Proportions of subjects who achieved complete wound closure by the classification of location of diabetic foot ulcer, Plantar and the other location between the two groups | During 12 weeks(at every visit during treatment period)
  Proportions of subjects who achieved complete wound closure
Durability of complete wound closure | Follow up to 24 weeks from the initial complete wound closure.
  Wound size is measured by using eKare 3D Wound Measurement system(Mobile Devices)

CONTACTS AND LOCATIONS:
Overall Officials: David G. Armstrong, MD.Ph D., Principal Investigator — University of Southern California; Alexander M. Reyzelman, DPM, Principal Investigator — Center for Clinical Research; Young Nathan, DPM, Principal Investigator — Martinsville Research Institute
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No